CLINICAL TRIAL: NCT06574867
Title: REQUEST - RemotE Monitoring by viQtor Upon Implementation on a Surgical departmenT
Brief Title: Evaluation of the viQtor Monitoring Solution on Surgical Wards
Acronym: REQUEST
Status: Recruiting | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Ephrahim Jerry, Drs., Catharina Ziekenhuis Eindhoven
Other Study IDs: NL. REQUEST
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Monitoring; Post-operative Monitoring; Patient Safety; Healthcare Technology Implementation; Contiuous Vital Signs Monitoring
Keywords: Continuous monitoring; Post-operative care; Vital signs; Healthcare technology; Wearable medical device; viQtor solution; Remote monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Patients Monitored with viQtor: This group includes adult patients admitted to the surgical ward at Catharina Hospital Eindhoven. Participants in this group will be monitored continuously using the viQtor wearable device to track vital signs such as heart rate, respiratory rate, and blood oxygen saturation during their hospital stay. The focus is on evaluating the implementation, usability, and effectiveness of the viQtor solution in a real-world clinical setting.
  Interventions: Device: viQtor Wearable Monitoring Device

INTERVENTIONS:
Device: viQtor Wearable Monitoring Device — The viQtor device is a wearable medical device designed for continuous monitoring of vital signs, including heart rate (PR), respiratory rate (RR), and blood oxygen saturation (SpO2). It is worn on the upper arm and transmits data wirelessly to a cloud-based platform. This device is being evaluated as part of the standard monitoring protocol for post-operative patients in a surgical ward setting.

SUMMARY:
The REQUEST study aims to evaluate the use of a new wireless monitoring device, called the viQtor solution, on a surgical ward in Catharina Hospital Eindhoven. This device continuously tracks vital signs, such as heart rate, breathing rate, and blood oxygen levels, in patients after surgery. The goal is to see if the viQtor solution can help detect health problems earlier and reduce the workload for nurses by minimizing the need for manual checks. The study will involve 500 patients and will take place over 7 months.

DETAILED DESCRIPTION:
Detailed Description

This is a prospective implementation evaluation study of the viQtor solution, a wearable medical device designed for continuous monitoring of vital signs in post-operative patients. The study will be conducted at the Catharina Hospital Eindhoven on the surgical ward "5 Oost" and will be divided into two phases, each involving approximately 250 patients.

In Phase 1 (Months 1-3), patients will continue to receive standard care, which includes manual spot checks and Modified Early Warning Score (MEWS) assessments by nursing staff. During this phase, healthcare professionals will receive training on how to use the viQtor solution.

In the Evaluation and Validation Period (Month 4), the accuracy of the viQtor device will be validated by comparing its continuous monitoring data with the manual measurements taken by nurses.

In Phase 2 (Months 5-7), the viQtor solution will become the primary method for monitoring patients, with manual checks conducted only when necessary. The study aims to assess the viQtor solution's usability, acceptance, adoption by healthcare professionals, and its accuracy in detecting patient deterioration. It will also evaluate the feasibility of implementing this technology in a real-world hospital setting and its impact on clinical outcomes.

The viQtor solution is a CE-marked Class IIa medical device, ensuring compliance with European safety standards. It is designed to be worn on the upper arm and is capable of wirelessly transmitting data every five minutes to a cloud-based platform accessible to healthcare professionals.

Participants in this study will include adult patients admitted to the surgical ward for various procedures. The study will not only assess the technical performance of the viQtor solution but also its impact on the workflow and workload of healthcare providers.

Data collected during the study will be used to determine the potential benefits and challenges of implementing continuous monitoring technology in hospital settings. The ultimate goal is to improve patient safety and outcomes through early detection of health deterioration, while also reducing the burden on nursing staff.

If successful, this study could pave the way for broader adoption of wearable monitoring technology in hospitals, potentially setting a new standard of care for post-operative patients.

This detailed description provides a comprehensive overview of the study objectives, methodology, and expected outcomes without duplicating information entered elsewhere in the record.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older).
* Patients admitted to the surgical ward at Catharina Hospital Eindhoven.
* Fluent in Dutch or English.
* Willingness to participate in the study and to wear the viQtor monitoring device during their hospital stay.

Exclusion Criteria:

Patients with cognitive impairments.

* Patients with allergies to metal or plastics.
* Patients with significant deformities, swelling, irritation, degenerative changes, or edema of the upper arm.
* Patients with implanted cardiac pacemakers, internal cardioverter defibrillators, or chronic resynchronization therapy devices.
* Patients at risk of vascular compromise of the arm on which the device will be placed.
* Patients with conditions that contraindicate the use of a blood pressure cuff or similar devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult post-operative patients admitted to the surgical ward at Catharina Hospital Eindhoven. The study will focus on evaluating the feasibility and effectiveness of continuous vital sign monitoring using the viQtor device.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Usability of the viQtor Monitoring Solution | 8 months
  Evaluation of the usability of the viQtor solution based on the System Usability Scale (SUS). The outcome will be measured by the SUS score, with a target score of >68 indicating acceptable usability.

SECONDARY OUTCOMES:
Reduction in Nursing Workload | 8 months
  Assessment of the reduction in nursing workload by comparing the time spent on manual spot checks before and after implementing the viQtor solution. Success is defined as a 20% reduction in time spent on manual checks.
Predictive Accuracy of the viQtor Solution | 8 months
  Evaluation of the viQtor solution's accuracy in predicting patient deterioration by comparing the continuous vital sign measurements (SpO2, PR, RR) with intermittent measurements conducted as part of the MEWS protocol.
Implementation Success of the viQtor Solution | 8 months
  Determination of the successful implementation of the viQtor solution, measured by the percentage of available and usable data (>70%) collected from the device during the study period.

OTHER OUTCOMES:
Nurse and Physician Adoption of the viQtor Solution | 8 months
  Measurement of the level of adoption and acceptance of the viQtor solution among healthcare staff, assessed through the Evidence-Based Practice Attitude Scale (EBPAS).

CONTACTS AND LOCATIONS:
Overall Officials: Simon S.W. Nienhuijs, Dr. PHD., Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns about patient privacy and confidentiality. The data collected includes sensitive health information, and sharing it could risk breaching participant anonymity. Additionally, the study's data use agreements and local regulations do not permit the sharing of IPD with external researchers.

REFERENCES:
- [Derived] Jerry EE, Bouwman AR, Nienhuijs SW. Remote Monitoring by ViQtor Upon Implementation on a Surgical Department (REQUEST-Trial): Protocol for a Prospective Implementation Study. JMIR Res Protoc. 2025 Jul 3;14:e70707. doi: 10.2196/70707. PMID 40608408